CLINICAL TRIAL: NCT05746962
Title: Safety and Efficacy of Colonoscopy Magnetic Imaging Device for Beginner Endoscopist: a Prospective Randomized Single-center Single-blind Study
Brief Title: Efficacy of Magnetic Imaging Colonoscopy Applied to Beginner Endoscopists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Keum, Bo Ra, Professor of Division of Gastroenterology and Hepatology, Department of Internal Medicine, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022AN0126
Record Dates: First submitted 2022-06-30; First posted 2023-02-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Colonic Neoplasms
Keywords: colonoscopy; loop formation; scopeguide
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group that does not use the scopeguide screen (Active Comparator): The control group should remove the looping of colonoscope by looking at the general colonoscopy screen The control group cannot use scopeguide screen Scopeguide screen is blinded by an opaque wrapping paper
  Interventions: Device: ScopeGuide Navigated Colonoscope
- Group using the scopeguide screen (Experimental): The experimental group uses a general endoscopic image during colonoscopic insertion The experimental group should remove the looping of colonoscope by looking at the scopeguide screen
  Interventions: Device: ScopeGuide Navigated Colonoscope; Device: Navigation screen

INTERVENTIONS:
Device: ScopeGuide Navigated Colonoscope — colonoscopes equipped with ScopeGuide
Device: Navigation screen — ScopeGuide's 3D visualisation screen
  Arms: Group using the scopeguide screen

SUMMARY:
Magnetic endoscopic imaging (scopeguide) is known to be helpful for colonoscope insertion, especially beginner endoscopist. In this trial, study was designed to show the efficacy and safety pertinent to scopeguide use in detail.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most commonly diagnosed malignancies worldwide. Colorectal cancer screening significantly reduced the incidence and mortality, and colonoscopy is generally recognized as a standard method. Among them, magnetic endoscopic imaging (MEI, Scopeguide, Magnetic Enhanced Instrument, Olympus, Japan) is a non-radiological imaging instrument that can display the three-dimensional configuration and position of the colonoscope in the abdominal cavity in real time. This study aims to investigate the effectiveness of colonoscopy by measuring the insertion-related index of the colonoscopy according to the scope guide for only beginners of endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age 19-80
* the patient who visit to examine the colonoscopy

Exclusion Criteria:

* the patient who has a pacemaker
* the patient who has electronic devices in the body
* bowel obstruction and bleeding
* glomerulus filter rate < 30
* inflammatory bowel disease, pregnancy
* previous history of bowel resection and abdominal surgery
* who refuse to write the informed consent
* previous history of allergic reaction to sedative drugs and beans, egg
* SBP <80, SpO2<90

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-08-28 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
proportion of colonoscope loop formation | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  proportion of colonoscope loop formation

SECONDARY OUTCOMES:
loop type | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  loop type
loop location | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  loop location
cecal intubation time cecal intubation time and rate | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  cecal intubation time
cecal intubation rate cecal intubation time and rate | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  success rate of cecal intubation
solving time for loop reduction | during colonoscope insertion, from the time that recognizes the loop and tries to resolve the looping of colonoscope to the time that completely resolved the colonoscope looping
  solving time for loop reduction
trial number of looping during loop reduction | during colonoscope insertion, the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  number of loop reduction trial
A method to eliminate the loop of colonoscope | during colonoscope insertion, the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  how to solve the looping of colonoscope, ex) clockwise rotation, anti-clockwise rotation
loop removal | during colonoscope insertion and after cecum arrival of colonoscope
  success or failure of loop removal
location of loop removal whether loop reduction success and location of loop reduction | during colonoscope insertion and after cecum arrival of colonoscope
  the colonic location where loop reduction success
total examination time | the time from the insertion of the colonoscope tip into the anal verge until withdrawal of the colonoscope from the cecum towards the anus
  total examination time
withdrawal time | the time during withdrawal of the colonoscope towards the anus
  withdrawal time (=examination time - cecal intubation time)
polyp detection rate | during whole colonoscopy examination
  polyp detection rate
adenoma detection rate | during whole colonoscopy examination
  adenoma detection rate
total sedation dose | during whole colonoscopy examination
  total sedation dose during colonoscopy
length of total inserted colonoscope | after arrival at the cecum
  length of total inserted colonoscope
application of pressure | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  nurse assissted abdominal pressure
patient position change | the time from the insertion of the colonoscope tip into the anal verge until reaching the cecum
  patient position change during colonoscope insertion
variance of blood pressure | during whole colonoscopy examination
  variance of blood pressure
variance of heart rate | during whole colonoscopy examination
  variance of heart rate
variance of respiration rate | during whole colonoscopy examination
  variance of respiration rate
variance of saturated oxygenation rate | during whole colonoscopy examination
  variance of saturated oxygenation rate
adverse events | during whole colonoscopy examination
  bleeding, perforation, and mucosal abrasion during colonoscopic exam
patients satisfaction (questionnaire) | during whole colonoscopy examination
  assessment for pain score through the examination
endoscopists satisfaction (questionnaire) | during whole colonoscopy examination
  assessment for maneuverability and difficulty score about insertion through the examination
evaluation of risk factors about loop formation | during whole colonoscopy examination
  factors that make a colonoscope loop

CONTACTS AND LOCATIONS:
Overall Officials: Bora Keum, Study Director — borakeum@hanmail.net
Locations (1):
- Han Jo Jeon, Seoul, Seong Buk Gu, South Korea